CLINICAL TRIAL: NCT07184879
Title: Comparison of Five Anesthetic Delivery Systems for Palatal Infiltration: A Randomized Clinical Trial
Brief Title: Comparison of Five Anesthetic Delivery Systems for Palatal Infiltration
Acronym: PAL-INJECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sercan Küçükkurt (Other)
Responsible Party: Sponsor-Investigator, Sercan Küçükkurt, Assoc. Prof. Dr. Sercan Küçükkurt, Oral and Maxillofacial Surgeon, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAU-PalatalRCT-2025
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Dental Anxiety; Pain; Dental; Palatal Anesthesia
Keywords: Dental Anesthesia; Palatal Infiltration; Visual Analog Scale (VAS); Computer-Controlled Local Anesthetic Delivery (CCLAD); Needle-Free Jet Injector; Injection Pain; Patient Fear; Dental Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-arm superiority clinical trial with five intervention groups comparing anesthetic delivery systems for palatal infiltration.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blind design: outcome assessors and the statistician were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Conventional Dental Syringe (CDS) (Experimental): Palatal infiltration using a conventional dental syringe with 27G needle; manual injection of 0.4 mL articaine with epinephrine over 15-20 seconds, with aspiration. Intervention Name: Device: Conventional Dental Syringe
  Interventions: Device: Conventional Dental Syringe
- Manual Pressure Syringe (MCJ) (Experimental): Palatal infiltration using ASPIJECT™ manual pressure syringe with 30G, 16 mm needle; manually controlled injection of 0.4 mL articaine with epinephrine over 15-20 seconds, with aspiration. Intervention Name: Device: Manual Pressure Syringe (ASPIJECT™)
  Interventions: Device: Manual Pressure Syringe (MCJ, ASPIJECT™)
- Spring-Activated Syringe (PCJ) (Experimental): Palatal infiltration using PAROJECT™ spring-activated syringe; two calibrated 0.2 mL doses of articaine with epinephrine following aspiration. Intervention Name: Device: Spring-Activated Syringe (PAROJECT™)
  Interventions: Device: Spring-Activated Syringe (PCJ, PAROJECT™)
- Needle-Free Jet Injector (NFI) (Experimental): Palatal infiltration using Comfort-in™ needle-free jet injector; 0.4 mL articaine with epinephrine delivered in <1 second, at 4-5 bar pressure; aspiration not applicable. Intervention Name: Device: Needle-Free Jet Injector (Comfort-in™)
  Interventions: Device: Needle-Free Jet Injector (NFI, Comfort-in™)
- Computer-Controlled Local Anesthetic Delivery (CCLAD) (Experimental): Palatal infiltration using CALAJECT™ Program I; 30G, 16 mm needle; AutoFlow delivery (0.006-0.009 mL/s) with automatic aspiration; microprocessor-controlled constant pressure. Intervention Name: Device: Computer-Controlled Local Anesthetic Delivery (CALAJECT™)
  Interventions: Device: Computer-Controlled Local Anesthetic Delivery (CCLAD, CALAJECT™)

INTERVENTIONS:
Device: Conventional Dental Syringe — Palatal infiltration anesthesia using a conventional dental syringe with a 27G needle. A total of 0.4 mL of articaine 4% with epinephrine 1:100,000 was administered manually over 15-20 seconds following aspiration.
  Arms: Conventional Dental Syringe (CDS)
Device: Spring-Activated Syringe (PCJ, PAROJECT™) — Palatal infiltration using a spring-activated push-button syringe (PAROJECT™). Two calibrated 0.2 mL doses of articaine 4% with epinephrine 1:100,000 were administered following aspiration.
  Arms: Spring-Activated Syringe (PCJ)
Device: Needle-Free Jet Injector (NFI, Comfort-in™) — Palatal infiltration using a needle-free jet injector (Comfort-in™). A total of 0.4 mL of articaine 4% with epinephrine 1:100,000 was delivered in less than one second at 4-5 bar pressure. Aspiration not applicable.
  Arms: Needle-Free Jet Injector (NFI)
Device: Computer-Controlled Local Anesthetic Delivery (CCLAD, CALAJECT™) — Palatal infiltration using a computer-controlled local anesthetic delivery system (CALAJECT™, Program I) with a 30G, 16 mm needle. AutoFlow rate 0.006-0.009 mL/s, with automatic aspiration after 5 seconds and constant microprocessor-controlled pressure. A total of 0.4 mL of articaine 4% with epinephrine 1:100,000 was administered.
  Arms: Computer-Controlled Local Anesthetic Delivery (CCLAD)
Device: Manual Pressure Syringe (MCJ, ASPIJECT™) — Palatal infiltration using a manual pressure-controlled syringe (ASPIJECT™) with a 30G, 16 mm needle. A total of 0.4 mL of articaine 4% with epinephrine 1:100,000 was administered manually over 15-20 seconds with aspiration.
  Arms: Manual Pressure Syringe (MCJ)

SUMMARY:
This study is a randomized clinical trial evaluating five different anesthetic delivery systems for palatal infiltration in adults undergoing maxillary molar extraction. A total of 200 healthy volunteers were enrolled and randomly assigned to receive anesthesia using one of the following devices: conventional dental syringe, manual pressure syringe, spring-activated syringe, needle-free jet injector, or computer-controlled local anesthetic delivery system.

The purpose of the study is to compare patient-reported pain, dental fear, and physiological responses (pulse rate and oxygen saturation) associated with each system. The results are expected to provide evidence on which devices may improve patient comfort and cooperation during palatal infiltration procedures.

DETAILED DESCRIPTION:
This randomized, parallel-arm superiority trial was conducted at Istanbul Aydın University, Faculty of Dentistry, between September 2023 and March 2025. Two hundred healthy adults (≥18 years) requiring maxillary molar extraction under palatal infiltration anesthesia were equally randomized into five groups (n=40).

All participants received 0.4 mL of 4% articaine with 1:100,000 epinephrine, delivered with one of the five systems. The primary outcome was pain perception measured immediately after injection using a visual analog scale (VAS). Secondary outcomes included changes in dental fear, pulse rate, oxygen saturation, and any adverse events.

The study was approved by the Istanbul Aydın University Ethics Committee. Written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA physical status I or II
* No systemic conditions affecting anesthetic metabolism
* No known allergy to local anesthetics or vasoconstrictors
* No psychiatric disorders or anxiolytic medication
* Ability to provide written informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Active infection at the injection site
* Diagnosed needle phobia
* Prior exposure to any of the tested injection systems
* Use of premedication, sedatives, or topical anesthetics on the day of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Pain during injection (VAS, 0-10 cm) | Immediately after injection
  Pain perception recorded immediately after palatal infiltration using a 10-cm visual analog scale (VAS; 0 = no pain, 10 = worst imaginable pain).

SECONDARY OUTCOMES:
Change in dental fear (VAS, 0-10 cm) | Baseline (before injection) and immediately after injection
  Fear measured on a 10-cm VAS before and after injection; difference (ΔVAS) represents fear reduction.
Pulse rate (bpm) | Baseline (before injection), peri-procedural (during injection), and 3 minutes post-injection
  Pulse rate measured with fingertip oximeter at three time points: baseline (before injection), peri-procedural (during injection), and 3 minutes after injection.
Oxygen saturation (SpO₂, %) | Baseline (before injection), peri-procedural (during injection), and 3 minutes post-injection
  Oxygen saturation measured with fingertip oximeter at three time points: baseline (before injection), peri-procedural (during injection), and 3 minutes after injection.
Adverse events | From the time of injection through study completion (average of 1 week follow-up)
  Recording of any immediate or delayed adverse events associated with anesthetic delivery (pain, swelling, bleeding, syncope, allergic reactions).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality and ethical restrictions. Aggregate results are available in the published manuscript.